CLINICAL TRIAL: NCT05135819
Title: Cyber School for Grandparents: an Intergenerational Educational Program to Bridge the Digital Divide
Brief Title: Cyber School for Grandparents: an Intergenerational Educational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Guaita, MD (Other)
Collaborators: University of Milano Bicocca (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor-Investigator, Antonio Guaita, MD, MD, Fondazione Golgi Cenci
Organization: Fondazione Golgi Cenci (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Intergenerational Relations; Aging Well
Keywords: Educational intervention; Digital divide; Social inclusion; Technology use; Old adults; Intergenerational relations; Learning
MeSH Terms: conditions — Social Inclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intergenerational educational program (Experimental)
  Interventions: Behavioral: Cyber School for Grandparents

INTERVENTIONS:
Behavioral: Cyber School for Grandparents — Educational program for secondary school students to become cyber tutors for their grandparents or for senior citizens, who are interested to learn new digital use and skills.

SUMMARY:
Social participation and social relationships are relevant aspects of older adult's psychosocial well-being. In this regard, specific interest is devoted to Information and Communication Technologies (ICT) which enable to connect people and to support their social participation.

Despite the number of older Internet users constantly increased in the last decades, older adults still display reduced Internet access compared to younger generations. Italian elderly people are severely penalized by this "gray digital divide". The pandemia due to COVID-19 spread has exasperated the situation, leading to the paradox of having people putatively most beneficent of use as those most excluded, due to scanty of competencies and of suitable and agreeable learning occasions.

The Cyber School for Grandparents is an innovative intergenerational educational program aimed to bridge the digital divide by training secondary school students (aged 15-17 years) to become cyber tutors for their grandparents.

The intervention will take place during the 2021/2022 school year, as part of the curricular activities of 3 classes at the local Human Science High School. The intervention was designed to be personalized and inclusive, in order to meet the need of each student-senior dyad, regardless of their starting digital skills and attitudes toward technology.

The primary aim of the present mixed-method feasibility study is to qualitatively evaluate students' participation and learning throughout the course and to measure grandparents' pre-post changes in mobile device actual use, self-reported proficiency and attitudes.

Secondly, eventual pre-post changes on aging stereotypes and psychosocial well-being of the participants will be explored.

DETAILED DESCRIPTION:
Systematic reviews of qualitative studies on older adults ICT users highlighted that the principal drives for use were the desire to keep in touch with family and friends and to enter into intergenerational communication, whereas main obstacles are their distrust in terms of perceived utility, privacy concerns as well as technical difficulties. As regards the learning context, old persons prefer to rely on their own social network to acquire digital competence and spontaneously refer to their younger family members that may act as "warm" experts on ICT use. ICT use among older adults may thus be favored by properly designed educational interventions, focused on their interests, needs and concerns about technology.

The educational program will be delivered to 3 classes of the local Human Science High School. Students will be asked to involve at least one grandparent willing to participate in the initiative. To assure the active participation of the entire classes, if some students were not able to involve any grandparent, community-dwelling older adults would be enrolled among those participating in ongoing studies at the Golgi Cenci Foundation.

Compared to the previously reported intergenerational programs on ICT use, the present initiative shows relevant innovative features: the educational lessons will be embedded in the students school program instead of being offered on a volunteering basis, the students will independently plan and implement the cyber sessions for their grandparents outside the school as extracurricular activities and, whenever possible, the program will involve familial dyads.

The course is composed of 3 different modules: theory (2 lessons), method (2 lessons) and practice (6 lessons). Theoretical lessons will deal with the aging process and its effect on cognition and learning process, issues and peculiarities of older adults ICT use, andragogy and strategies to favor the learning process of new skills.

During the methodological lessons, students will be instructed on the importance of data collection for research purposes and on the specific features and administration modalities of the assessment tools to be compiled by their grandparents.

In the practical module, students will be guided in the implementation of the one-to-one cyber sessions for their grandparents, which will be then conducted independently during extracurricular hours and customized according to the needs and interests of each senior involved.

Pre-post outcome measures will be remotely collected both for students and for seniors. Assessment will be performed through online surveys shared within the web-based platform adopted by the school to perform remote lessons during the COVID-19 pandemic (Google Classroom). All the instruments selected are suitable for self-compiling both by young students and older adults. The students will help and supervise grandparents to manage possible technical and/or sensory difficulties with the online compiling procedure.

Moreover, students will compile an online diary for each of the 4 practical modules, before the next group lesson scheduled, comprising both an activity and a learning log. The activity log consists of structured questions on the number, frequency, duration, content and modality (in-person or remotely) of the cyber sessions performed with the senior mentee. The learning log will comprise broad guiding questions to reflect on the learning process favoured by the activities and to record the student's observations.

Finally, at the end of the experience, students and grandparents satisfaction and opinion on the experience will be assessed using a questionnaire with both close-ended and open-ended questions.

ELIGIBILITY:
Inclusion criteria:

* For students: attending one of the 3 classes involved in the project
* For seniors: be a grandparents of the students involved and willing to participate in the initiative.

No specific inclusion criteria were set regarding age, ICT proficiency, socioeconomic, health or mobility status of the grandparents, since the program was expressly designed to be as inclusive and personalized as possible, in order to favor a wide participation.

However, context information on these relevant aspects will be collected and reported, since they are well-known factors affecting technology use among older adults.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Digital literacy (seniors) | 5 months
  Mobile Device Proficiency Questionnaire Short Form (MDPQ-SF): self report, 16 items on the 5 dimensions of the European digital competence framework evaluated on a 5-point Likert scale (range: 16-80)
Attitude toward Internet use (seniors) | 5 months
  Attitude Toward Computer/Internet Use Questionnaire (ATCQ): self report, 15 items measuring 5 attitude dimensions (comfort, efficacy, interest) toward Internet use on a 5-point Likert scale (range: 15-75)

SECONDARY OUTCOMES:
Psychosocial well-being (students and seniors) | 6 months
  Mental Health Continuum Short Form (MHC-SF): self report, 14 item measuring 3 dimension of well-being (emotional, social, psychological) on a 6-point Likert scale (range: 0-70)
Aging stereotype (students) | 6 months
  Aging semantic differential: 9 pairs of polar opposite adjectives on aging individuals, to rate the intensity and direction of judgement from 0 to 7.

OTHER OUTCOMES:
Students participation | 4 months
  Number of the cyber sessions organized with the senior, reported by students on the online diary (activity log)
Students learning | 4 months
  Qualitative evaluations of the responses to open-ended questions on the online diary (learning log)
Seniors mobile device actual use changes | 4 months
  Analysis of log data recorded by a specific app installed on the device (Rescue Time)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Rolandi, MSc, Principal Investigator — Fondazione Golgi Cenci
Locations (1):
- Golgi Cenci Foundation, Abbiategrasso, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nef T, Ganea RL, Muri RM, Mosimann UP. Social networking sites and older users - a systematic review. Int Psychogeriatr. 2013 Jul;25(7):1041-53. doi: 10.1017/S1041610213000355. Epub 2013 Apr 4. PMID 23552297
- [Background] Ibarra F, Baez M, Cernuzzi L, Casati F. A Systematic Review on Technology-Supported Interventions to Improve Old-Age Social Wellbeing: Loneliness, Social Isolation, and Connectedness. J Healthc Eng. 2020 Jul 12;2020:2036842. doi: 10.1155/2020/2036842. eCollection 2020. PMID 32765823
- [Background] Forsman AK, Nordmyr J, Matosevic T, Park AL, Wahlbeck K, McDaid D. Promoting mental wellbeing among older people: technology-based interventions. Health Promot Int. 2018 Dec 1;33(6):1042-1054. doi: 10.1093/heapro/dax047. PMID 28973587
- [Background] Roque NA, Boot WR. A New Tool for Assessing Mobile Device Proficiency in Older Adults: The Mobile Device Proficiency Questionnaire. J Appl Gerontol. 2018 Feb;37(2):131-156. doi: 10.1177/0733464816642582. Epub 2016 Apr 11. PMID 27255686
- [Background] Rolandi E, Vaccaro R, Abbondanza S, Casanova G, Pettinato L, Colombo M, Guaita A. Loneliness and Social Engagement in Older Adults Based in Lombardy during the COVID-19 Lockdown: The Long-Term Effects of a Course on Social Networking Sites Use. Int J Environ Res Public Health. 2020 Oct 28;17(21):7912. doi: 10.3390/ijerph17217912. PMID 33126634
- [Background] Jay GM, Willis SL. Influence of direct computer experience on older adults' attitudes toward computers. J Gerontol. 1992 Jul;47(4):P250-7. doi: 10.1093/geronj/47.4.p250. PMID 1624702
- [Background] Keyes CL. The mental health continuum: from languishing to flourishing in life. J Health Soc Behav. 2002 Jun;43(2):207-22. PMID 12096700